CLINICAL TRIAL: NCT00844181
Title: Racial Differences in Orthostatic Tolerance
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Nina Stachenfeld, PhD, John B. Pierce Laboratory
Other Study IDs: 0512000875; 3R01HL071159-04A1S1 (NIH)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Orthostatic Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 0: white women
- 1: Black women

SUMMARY:
Our central hypothesis is that baroreflex sensitivity is attenuated in black women compared to white women, and that this dysregulation will be apparent during orthostatic challenges. We expect that the cumulative stress index (CSI), a measure of maximal orthostatic tolerance, is higher in Black women (BW) compared to White women (WW).

ELIGIBILITY:
Inclusion Criteria:

* women between 18-25 yrs of age

Exclusion Criteria:

* history of high blood pressure, uterine fibroids, diabetes, epilepsy

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of women of reproductive age
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
orthostatic tolerance | 1

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, PhD, Principal Investigator — Yale University
Locations (1):
- John B. Pierce Laboratory, New Haven, Connecticut, United States